CLINICAL TRIAL: NCT06470750
Title: Feasibility of Patient-Centered Home Care (PCHC) to Reduce Disparities in High-Risk Black Men (BM) With Advanced Prostate Cancer (CaP)
Brief Title: Feasibility of Patient-Centered Home Care (PCHC) to Reduce Disparities in High-Risk Black Men (BM) With Prostate Cancer (CaP)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: CaP PCHC; W81XWH2210969 (Other Grant/Funding Number: Department of Defense); W81XWH2210968 (Other Grant/Funding Number: Department of Defense); NCI-2024-04792 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 22-004375 (Other: Mayo Clinic Institutional Review Board); CaP PCHC (Other: Mayo Clinic in Florida)
Record Dates: First submitted 2024-06-18; First posted 2024-06-24 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Prostate Adenocarcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Observational group 1: Participants take part in a focus group or complete questionnaires and may take part in an interview on study.
  Interventions: Other: Non-Interventional Study
- Observational group 2: Participants complete questionnaires throughout the study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study evaluates the possibility of patient-centered home care as a new model of cancer care to reduce disparities and improve health related quality of life and patient-reported outcomes in Black patients with prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To evaluate a highly innovative project evaluating the feasibility of patient-centered home care PCHC as a new model of cancer care to reduce disparities and improve health related QoL (HRQoL) and patient reported-outcomes (PROs) in Black patients with advanced prostate cancer (CaP). (Phase I) II. Establish patient-centeredness by exploring patients' choice relative to the place of CaP treatment for certain aspects of therapy as well as end-of-life care.

III. Establish the acceptance and impact of PCHC on PROs and HRQoL in BM with advanced CaP.

OUTLINE: This is an observational study. Participants are assigned to 1 of 2 groups.

GROUP 1: Participants take part in a focus group or complete questionnaires and may take part in an interview on study.

GROUP 2: Participants complete questionnaires throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* GROUP 1 FOCUS GROUPS:

  * Individuals identifying as Black and male who are familiar with the landscape of medical care and cancer
* GROUP 1 SURVEYS:

  * Are 18 years of age or older
  * Have histologic evidence of prostate adenocarcinoma
  * Are requiring, have required, or will require prostate cancer treatment
  * Have an understanding of the protocol and its requirements
  * Are willing to fill in a questionnaire and participate in a focused interview
  * Are able and willing to sign an informed consent
* GROUP 1 INTERVIEWS:

  * Enrollment in the survey phase of the protocol
* GROUP 2:

  * Are 18 years of age or older
  * Are Black men or other discounted patients (older adults, individuals residing in rural or remote areas, and those facing transportation challenges)
  * Have histologic evidence of prostate adenocarcinoma
  * Are requiring active standard hormone-based therapies (degarelix or leuprolide), antibone resorptive agents (zoledronic acid or denosumab), oral anticancer treatments (abiraterone or second-generation androgen receptor blockers) or intravenous chemotherapy (docetaxel)
  * Are receiving part of supportive care/symptom management and/or anti-cancer therapy in the home as part of Cancer Care Beyond Walls (CCBW)
  * Have an understanding of the protocol and its requirements
  * Are able and willing to sign informed consent

Exclusion Criteria:

* GROUP 1 FOCUS GROUPS:

  * Individuals who do not identify as Black or male or who have had no extensive interaction with the healthcare system
* GROUP 1 SURVEYS:

  * Do not identify as Black men
  * Have not been diagnosed with prostate cancer
* GROUP 1 INTERVIEWS:

  * Not enrolled in the survey phase of the protocol
* GROUP 2:

  * Do not identify as Black men or other discounted patients (older adults, individuals residing in rural or remote areas, and those facing transportation challenges)
  * Have not been diagnosed with histologic evidence of prostate adenocarcinoma
  * Are not requiring active standard anti-cancer therapy

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Individuals identifying as Black and male who are familiar with the landscape of medical care and cancer, as well as individuals identifying as an African American/Black man with prostate adenocarcinoma requiring prostate cancer therapy and individuals identifying as an African American/Black man with prostate adenocarcinoma requiring active standard hormone-based therapies, antibone resorptive agents, oral anticancer treatments, or intravenous chemotherapy and receiving part of supportive care/symptom management and/or anti-cancer therapy in the home as part of the Advanced Care at Home Program
Sampling Method: Non-Probability Sample
Enrollment: 77 (Estimated)
Dates: Start 2024-07-25 (Actual); Primary Completion 2026-07-30 (Estimated); Study Completion 2026-07-30 (Estimated)

PRIMARY OUTCOMES:
Feasibility of Patient-centered Home Care (PCHC) | Up to 6 months
  Participants will be asked to fill in a brief questionnaire regarding: patient preference for location of therapy (at the infusion center or in the home); perceived difficulties (isolation, less contact with hospital staff and other patients, feeling less secure with less back-up outside the hospital setting, the possibility of equipment malfunctions and complications in the home setting); and advantages (less travelling to specialized medical facilities, reduced risk of hospital acquired infections or blood clots, the ability to receive treatment in the comfort and security of the home, less disruption to family life, increased feeling of control over treatment and illness). Feasibility will be assessed based on responses to the questionnaire.

SECONDARY OUTCOMES:
Time to emergency room visit | Up to 6 months
  Time to first emergency room visit will be recorded.
Time to hospital visit | Up to 6 months
  The time to first hospitalization will be recorded.

CONTACTS AND LOCATIONS:
Overall Officials: Roxana S. Dronca, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Florida, Jacksonville, Florida, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials